CLINICAL TRIAL: NCT02796261
Title: A Randomized Phase 3 Open-Label Study To Evaluate the Efficacy and Safety of Eflornithine With Lomustine Compared to Lomustine Alone in Patients With AA That Progress/Recur After Irradiation and Adjuvant Temozolomide Chemotherapy
Brief Title: Study to Evaluate Eflornithine + Lomustine vs Lomustine in Recurrent Anaplastic Astrocytoma (AA) Patients
Acronym: STELLAR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Orbus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OT-15-001
Record Dates: First submitted 2016-06-03; First posted 2016-06-10 (Estimated); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Anaplastic Astrocytoma; Recurrent Anaplastic Astrocytoma
Keywords: Anaplastic Astrocytoma; Grade 3 Glioma; Glioma; Eflornithine; Brain Cancer; Brain Tumor; Neuro-oncology; Progressive Anaplastic Astrocytoma; Recurrent Anaplastic Astrocytoma; Progressive Glioma; Recurrent Glioma; Malignant Glioma; Progressive Brain Tumor; Recurrent Brain Tumor
MeSH Terms: conditions — Astrocytoma; Glioma; Brain Neoplasms | interventions — Eflornithine; Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eflornithine + Lomustine (Experimental): Eflornithine dosed on a 2 weeks on, 1 week off schedule + Lomustine dosed every 6 weeks
  Interventions: Drug: Eflornithine; Drug: Lomustine
- Lomustine (Active Comparator): Lomustine dosed every 6 weeks
  Interventions: Drug: Lomustine

INTERVENTIONS:
Drug: Eflornithine — Eflornithine 2.8 g/m2 administered orally every 8 hours on a 2 week on, 1 week off schedule
  Other Names: DFMO
  Arms: Eflornithine + Lomustine
Drug: Lomustine — Lomustine 90 mg/m2 administered orally once every 6 weeks
  Other Names: CCNU; CeeNU; Gleostine
  Arms: Eflornithine + Lomustine
Drug: Lomustine — Lomustine 110 mg/m2 administered orally once every 6 weeks
  Other Names: CCNU; CeeNU; Gleostine
  Arms: Lomustine

SUMMARY:
The purpose of this study is to compare the efficacy and safety of eflornithine in combination with lomustine, compared to lomustine taken alone, in treating patients whose anaplastic astrocytoma has recurred/progressed after radiation and temozolomide chemotherapy.

DETAILED DESCRIPTION:
This study will consist of 4 study periods of up to 50 months in total, consisting of:

Screening Period - A maximum screening duration of 4 weeks.

Treatment Period - Treatment Arm A up to 24 months; Treatment Arm B up to 12 months.

End of Treatment Visit - A minimum of 4 weeks post last treatment for both arms.

Follow-Up Period - Up to approximately 36 months, or until patient death.

A total of approximately 340 patients will be randomized in a 1:1 ratio to receive either eflornithine + lomustine or lomustine alone.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for participation in this study:

* Surgical or biopsy-proven diagnosis of WHO grade 3 AA.
* First AA tumor progression or recurrence ≤ 6 months prior to randomization based on MRI using T2 hyperintesity, gadolinium (Gd)-contrast enhancement, or both. To avoid enrollment of patients with glioblastoma, patients with Gd-contrast enhancing tumors will be eligible if there is no necrosis seen on MRI and any of the following criteria is true:

  1. Gd-contrast lesion margins are not clearly defined,
  2. Gd-contrast lesions are only measurable in one dimension,
  3. Gd-contrast lesion has two perpendicular diameters less than 10 mm,
  4. Gd-contrast lesion has two perpendicular diameters greater than 10 mm but less than 20 mm and lesion does not demonstrate central necrosis,
  5. Recent histopathological confirmation of WHO grade 3 AA
* Received EBRT and temozolomide chemotherapy prior to first tumor progression or recurrence of WHO Grade 3 AA.
* Completion of EBRT ≥ 6 months prior to randomization.
* A patient whose AA tumor has progressed or recurred and has had another surgical resection prior to randomization will be eligible if a) pathology review confirms AA, and b) post-surgical MRI demonstrates measurable tumor on T2 FLAIR.
* Karnofsky Performance Status (KPS) score of ≥ 70.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria are not eligible for study participation:

* MRI defining progression is consistent with a diagnosis of glioblastoma or radiation necrosis.
* Patients who are considered to be refractory to EBRT and temozolomide but who have not progressed.
* Prior systemic therapy for recurrence of AA.
* Presence of extracranial or leptomeningeal disease.
* Prior lomustine use.
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the patient unsuitable for the study.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2016-07; Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 4 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 4 years
Objective response rate (ORR) | 4 years

OTHER OUTCOMES:
Clinical benefit response (CBR) based on magnetic resonance imaging (MRI) criteria | 4 years
OS rate at 18 months (OS-18) | 18 months
Relevance of OS, PFS, ORR, and CBR to commonly used molecular/genetic biomarkers obtained from most recent pre-study tumor samples | 4 years
Pharmacokinetic Analysis - Maximum concentrations (Cmax) of eflornithine in plasma will be determined. | 1 Month
PK - Area under the curve (AUC) of eflornithine in plasma will be determined. | 1 Month

CONTACTS AND LOCATIONS:
Locations (79):
- United States (47):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Kaiser Permanente, Los Angeles, California
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - Kaiser Permanente Center, Redwood City, California
  - Kaiser Permanente, Sacramento, California
  - UCSD Moores Cancer Center, San Diego, California
  - University of California San Francisco Medical Center, San Francisco, California
  - John Wayne Cancer Institute, Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - University of South Florida (USF) - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Piedmont Physicians Neuro-Oncology, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Northwestern Medicine CDH Cancer Center, Warrenville, Illinois
  - The University of Iowa, Iowa City, Iowa
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Norton Cancer Institute - Louisville, Louisville, Kentucky
  - Louisiana State University Health Sciences Center New Orleans, New Orleans, Louisiana
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - HCA Midwest Division, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - JFK Medical Center, Edison, New Jersey
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center, The Neurological Institute, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Cleveland Clinic, Richard E. Jacobs Health Center, Cleveland, Ohio
  - OhioHealth Research and Innovation Institute, Columbus, Ohio
  - Providence Brain & Spine Institute, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Hollings Cancer Center, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Texas Oncology Austin Brain Tumor Center, Austin, Texas
  - Neuro-Oncology Associates, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Swedish Health Services, Seattle, Washington
- Belgium (2):
  - Universitair Ziekenhuis Leuven, Leuven, Flemish Brabant
  - Cliniques Universitaires UCL De Mont-Godinne, Yvoir, Namur
- Canada (6):
  - Tom Baker Cancer Center, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- France (8):
  - Institut de Cancerologie de l'Ouest - Angers, Angers
  - CHRU de Brest, Brest
  - Hôpital Pierre Wertheimer - Hospices Civils de Lyon, Bron
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Hôpital Roger Salengro, Lille
  - Hôpital de la Timone, Marseille
  - Hôpital Universitaire Pitié Salpêtrière, Paris
- Germany (4):
  - Klinik und Poliklinik fur Neurologie der Universitat Regensburg, Regensburg, Bavaria
  - Heinrich-Heine-Universitat Duesseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- Italy (3):
  - Fondazione IRCCS - Instituto Neurologico Carlo Besta, Milan
  - Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino - Ospedale Molinette, Torino
- Netherlands (4):
  - Sint Elisabeth Ziekenhuis, Tilburg, North Brabant
  - Vrije Universiteit Medisch Centrum (VUMC), Amsterdam, North Holland
  - Erasmus Medisch Centrum Daniel den Hoed, Rotterdam, South Holland
  - Universitair Medisch Centrum Utrecht, Utrecht
- United Kingdom (5):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Edinburgh Cancer Centre - Western General Hospital, Edinburgh
  - Guy's Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colman H, Lombardi G, Wong ET, Walbert T, Eoli M, Lassman AB, Peereboom DM, Kizilbash SH, Kamiya-Matsuoka C, Pitz MW, Strowd RE, Desjardins A, Kumthekar P, Mason W, Pellerino A, Soffietti R, Butowski N, Forsyth PA, Hamza MA, Hau P, Lallana E, Nabors B, Piccioni D, Uhlmann EJ, Welsh LC, Wen PY, Dietrich J, Wang C, Levin VA. STELLAR: Phase III, Randomized, Open-Label Study of Eflornithine Plus Lomustine Versus Lomustine Alone in Patients With Recurrent Grade 3 Astrocytoma. J Clin Oncol. 2025 Dec 1:JCO2501204. doi: 10.1200/JCO-25-01204. Online ahead of print. PMID 41325560